CLINICAL TRIAL: NCT04919980
Title: TVMR With the INNOVALVE System Trial - Early Feasibility Study
Acronym: TWIST-EFS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-13
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Mitral Valve Regurgitation (Degenerative or Functional)
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (Experimental): MV replacement with INNOVALVE system
  Interventions: Device: INNOVALVE system

INTERVENTIONS:
Device: INNOVALVE system — INNOVALVE system

SUMMARY:
Study to evaluate the safety and performance of the INNOVALVE system

DETAILED DESCRIPTION:
The study is a multi-center, First-In-Human, prospective, single arm early feasibility study to evaluate the safety and performance of the INNOVALVE system

ELIGIBILITY:
Inclusion Criteria:

* Clinically significant, symptomatic mitral regurgitation
* High risk for open-heart surgery
* Meets anatomical criteria

Exclusion Criteria:

* Unsuitable anatomy
* Patient is inoperable
* EF<25%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2031-07-01 (Estimated)

PRIMARY OUTCOMES:
Absence of implant or delivery related serious adverse events at 30 Days | 30 days
  Absence of implant or delivery related serious adverse events

SECONDARY OUTCOMES:
Technical success | Procedure
Procedural success | 30 days
NYHA functional class | 30 days, 6, 12 months and annually up to 5 years
Six-minute walk test | 30 days, 6, 12 months and annually up to 5 years
Quality of life improvement (KCCQ-12) | 30 days, 6, 12 months and annually up to 5 years
Reduction in MR grade | 30 days, 6, 12 months and annually up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Chet Rihal, Principal Investigator — Mayo Clinic
Locations (17):
- United States (17):
  - Cedars-Sinai, Los Angeles, California
  - Naples Comprehensive Health, Naples, Florida
  - Piedmont Heart Institute, Atlanta, Georgia
  - Northwestern, Chicago, Illinois
  - University of Michigan Hospital and Health Systems, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - Northwell Health, Manhasset, New York
  - Cornell, New York, New York
  - NewYork-Presbyterian / Columbia University, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - OhioHealth Research Institute, Columbus, Ohio
  - Oregon Health & Science Universtiy, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Ascension Saint Thomas, Nashville, Tennessee
  - Swedish Medical Center, Seattle, Washington